CLINICAL TRIAL: NCT05943847
Title: Evaluation of Neurotrophic Growth Factors in Breast Milk at Two Years of Age and Beyond
Brief Title: Neurotrophic Growth Factors in Breast Milk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Gonca Keskindemirci, Assoc Prof, Istanbul University
Other Study IDs: TSA-2023-39668
Record Dates: First submitted 2023-04-11; First posted 2023-07-13 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Breast Milk Collection
Keywords: Breast milk; BDNF; GDNF; S100B
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Breast milk will be stored due to analysis at 12th months of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to demonstrate the presence of neurotrophic factors in the breast milk of mothers with 18-month-old children and the persistence of these factors in breast milk after the age of 2 years. The main questions it aims to answer are:

* Does the breast milk of mothers with 18-month-old babies contain Brain-Derived Neurotrophic Factor (BDNF), S100B protein and glial cell line-derived neurotrophic factor (GDNF)?
* Does the breast milk continue to contain BDNF, s100B protein and GDNF and-after 24 months?

Participants will be asked to give breastmilk at 3 separate times. Breast milk samples will be collected from mothers at 18th-month, 24th-month and ≥25 months of their babies. A total of 75 breast milk samples obtained from 25 mothers with their consent will be analyzed.

DETAILED DESCRIPTION:
Growth factors are among the bioactive compounds found in breast milk and have effects on the growth and maturation of the baby's organs and systems. The completion of each organ maturation occurs at different times. Although the development of the nervous system reaches 60% of adults at the age of 2 years, it continues after the age of 2. Brain-Derived Neurotrophic Factor (BDNF), S100B protein, and glial cell line-derived neurotrophic factor (GDNF) are the neurotrophic growth factors found in breast milk and play a critical role in the development of the nervous system, the maintenance of neuronal functionality and the proliferation of neurons . They play a role during brain development, particularly in differentiating neuronal and glial cells. In addition, it is effective in synaptic plasticity and has important roles in the mature nervous system. The presence of neurotrophic factors in breast milk under the age of one has been demonstrated. However, the presence of these factors in breast milk has not been evaluated at 2 years and above. In this study, investigators aimed to demonstrate the presence of neurotrophic factors in the breast milk of mothers with 18-month-old children and the persistence of these factors in breast milk after the age of 2 years.

Study Design:

The study was conducted at Istanbul University, Istanbul Medical Faculty, Department of Pediatrics, Department of Social Pediatrics, Well Child Outpatient Clinic. All mothers participating in the study are informed in detail about the study and the importance of breast milk. According to Turkish Demographic and Health Survey (TDHS) 2018 data, the rate of breastfeeding is 66% at 12 months, 50% at 18 months, and 34% at 24 months. Considering the decrease according to age, it was assumed that the breastfeeding rate would be 18% after the age of 2. Considering the TDHS 2018 data of mothers, assuming that 18% of mothers breastfeed their babies after the age of 2, with a 95% confidence level and an acceptable sampling error of 0.15, the sample size calculation formula was used to estimate the population ratio, and the sample size was calculated for each mother. It is planned to have at least 25 mothers during the milk collection period (for each mother 18., 24., ≥ 25 months), with a total of 75 breast milk.

Breast milk collections and analysis:

1. Breast milk will be collected at 3 separate times at 18th-month, 24th-month and ≥25 months of their babies.
2. Using the manual milking method, 5 ml of expressed breast milk will be collected in Eppendorf tubes and transported in a polystyrene box containing ice (at 4°C) to the laboratory within 30 minutes. All breast milk samples will be stored at -20°C under laboratory conditions until the analysis.
3. All collected breast milk samples will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degrees one day before analysis, room temperature on the day of analysis) at the 12th month of the study. The neurotrophic factors (BDNF, S100B, GDNF) will be analyzed with ELISA (Elabsicence; United States) method.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who applied for the 18th-month follow-up of their exclusively breastfed baby for the first 6 months agreed to participate in the study.

Exclusion Criteria:

* Mothers of infants who were not exclusively breastfed in the first six months
* Mothers with infection, metabolic disease, central nervous system, breast disease or pregnancy
* Mothers of infants with infection, metabolic disease, malnutrition and central nervous system disease
* Mothers who stop breastfeeding before 25 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers will included
Study Population: On the basis of the inclusion and exclusion criteria 25 mothers will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2024-03-25 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of BDNF in the breastmilk at 18 months | Sample collection: 1-3 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected at the 18th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for BDNF with ELISA (E-lab-science; United States) method.
Analysis of BDNF in the breastmilk at 24 months months | Sample collection: 7-9 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected at the 24th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for BDNF with ELISA (E-lab-science; United States) method.
Analysis of BDNF in the breastmilk at ≥25 months | Sample collection: 8-11 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected after 24th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for BDNF with ELISA (E-lab-science; United States) method.
Analysis of GDNF in the breastmilk at 18 months | Sample collection: 1-3 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected at the 18th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for GDNF with ELISA (E-lab-science; United States) method.
Analysis of GDNF in the breastmilk at 24 months | Sample collection: 7-9 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected at the 24th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for GDNF with ELISA (E-lab-science; United States) method.
Analysis of GDNF in the breastmilk at ≥25 months | Sample collection: 8-11 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected after 24th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for GDNF with ELISA (E-lab-science; United States) method.
Analysis of S100B in the breastmilk at 18 months | Sample collection: 1-3 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected at the 18th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for S100B with ELISA (E-lab-science; United States) method.
Analysis of S100B in the breastmilk at 24 months | Sample collection: 7-9 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected at the 24th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for S100B with ELISA (E-lab-science; United States) method.
Analysis of S100B in the breastmilk at ≥25 months | Sample collection: 8-11 months of the study ; Analyze: 12th month of the study
  Breast milk samples which were collected after 24th month of the babies and stored in Eppendorf tubes at -20°C will be prepared for analysis by gradual thawing (breast milk will be taken to +4 C degree the day before analysis, room temperature on the day of analysis) in the 12th month of the study and will be analysed for S100B with ELISA (E-lab-science; United States) method.

SECONDARY OUTCOMES:
Sociodemographic factors | at the beginning (18. months of age)
  Maternal age, number of pregnancies, number of births
Maternal disease | at the beginning (18. months of age)
  Rate of mothers' diseases other than exclusion criteria, if any
Maternal drug use | at the beginning (18. months of age)
  Rate of medications used by mothers, if any

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Keskindemirci, Assoc Prof, Study Director — İstanbul Univeristy; Öykü Özbörü Aşkan, PhD, Principal Investigator — İstanbul Univeristy; Gülbin Gökçay, Prof, Principal Investigator — İstanbul Univeristy; Tülin Özden, Prof, Principal Investigator — İstanbul Univeristy; Alev Bakır Kayı, PhD, Principal Investigator — İstanbul Univeristy
Locations (1):
- İstanbul University İstanbul Medical Faculty Department of Pediatrics Division of Social Pediatrics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The decision will be made after the permission of the authors and authors' institution